CLINICAL TRIAL: NCT05973097
Title: Clinical Study of Combined Treatment of Oral Lichen Planus With Paeoniflorin and Photodynamic Therapy
Brief Title: Treatment of Oral Lichen Planus With Paeoniflorin and Photodynamic Therapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PUTHM912068
Record Dates: First submitted 2023-07-15; First posted 2023-08-02 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-07

CONDITIONS: Oral Lichen Planus
Keywords: oral lichen planus; integrated Chinese and Western medicine; total glucosides of paeony; photodynamic therapy
MeSH Terms: conditions — Lichen Planus, Oral

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- total glucosides of paeony treatment (Active Comparator): Total glucosides of paeony capsules were given 0.6 g once, 3 times a day.
  Interventions: Drug: total glucosides of paeony treatment
- photodynamic therapy treatment (Active Comparator): Cover the lesion with photosensitizer and fix it. Remove the photosensitizer and treat with laser diode.
  Interventions: Other: photodynamic therapy treatment
- glucosides of paeony and photodynamic therapy combined treatment (Experimental): Glucosides of paeony and photodynamic therapy are combined for the treatment
  Interventions: Other: glucosides of paeony and photodynamic therapy combined treatment

INTERVENTIONS:
Drug: total glucosides of paeony treatment — Total glucosides of paeony capsules were given 0.6 g once, 3 times a day.
  Arms: total glucosides of paeony treatment
Other: photodynamic therapy treatment — Cover the lesion with photosensitizer and fix it. Remove the photosensitizer and treat with laser diode.
  Arms: photodynamic therapy treatment
Other: glucosides of paeony and photodynamic therapy combined treatment — Glucosides of paeony and photodynamic therapy are combined for the treatment
  Arms: glucosides of paeony and photodynamic therapy combined treatment

SUMMARY:
Oral lichen planus (OLP) is a common chronic inflammatory disease of the oral mucosa and is considered a precancerous condition. It is characterized by white reticular changes in the oral mucosa, which can progress to erosions and cause pain in severe cases. The pathogenesis of OLP is still unclear, but it is believed to be a T-lymphocyte-mediated autoimmune disease. Currently, only symptomatic treatments are available, and there is no definitive cure.

In this project, we plan to use TCM differentiation to categorize OLP patients and conduct a randomized controlled clinical trial to demonstrate the enhanced therapeutic effect of paeoniflorin combined with photodynamic therapy for OLP. The implementation of this project will provide new insights into the clinical management of OLP, improve our understanding of the treatment mechanisms, and have important theoretical and clinical implications.

DETAILED DESCRIPTION:
Paeoniflorin, a compound extracted from the traditional Chinese medicine, has anti-inflammatory and immunomodulatory effects. Photodynamic therapy is a novel local treatment approach, where photosensitizers selectively target and destroy diseased cells. Both treatments have shown efficacy in treating OLP when used individually.

ELIGIBILITY:
Inclusion Criteria:

* patients with oral lichen planus
* male or female patients older than 18 years of age
* patients willing to participate with signed informed consent.

Exclusion Criteria:

* pregnant or lactating
* had serious systemic diseases of the heart, lung, liver, and kidney, or had tumors
* were unwilling to participate in the experiment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2023-07-30 (Estimated); Primary Completion 2028-12-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Efficacy at 1 month of treatment | 1 month
  According to the trial standard for evaluating the efficacy of atrophic and erosive oral lichen planus (OLP), the evaluation includes both objective and subjective measures.
  Objective measure: The size of the lesion is measured by an observer. The physician records and takes photographs of the lesion, noting the location, color, and changes in the area. The color and area changes of the lesion are compared and determined based on the photographic records.
  Subjective measure: Visual analogue scales (VAS) are used, which consist of 10 levels. The pain level is recorded, and the assessment is done by the patient.

SECONDARY OUTCOMES:
The curative effect at the later follow-up visit | through study completion, an average of 1 year
  According to the trial standard for evaluating the efficacy of atrophic and erosive oral lichen planus (OLP), the evaluation includes both objective and subjective measures.
  Objective measure: The size of the lesion is measured by an observer. The physician records and takes photographs of the lesion, noting the location, color, and changes in the area. The color and area changes of the lesion are compared and determined based on the photographic records.
  Subjective measure: Visual analogue scales (VAS) are used, which consist of 10 levels. The pain level is recorded, and the assessment is done by the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Zhihui Zhang, Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] van der Meij EH, van der Waal I. Lack of clinicopathologic correlation in the diagnosis of oral lichen planus based on the presently available diagnostic criteria and suggestions for modifications. J Oral Pathol Med. 2003 Oct;32(9):507-12. doi: 10.1034/j.1600-0714.2003.00125.x. PMID 12969224
- [Background] Li J, Chen CX, Shen YH. Effects of total glucosides from paeony (Paeonia lactiflora Pall) roots on experimental atherosclerosis in rats. J Ethnopharmacol. 2011 May 17;135(2):469-75. doi: 10.1016/j.jep.2011.03.045. Epub 2011 Mar 29. PMID 21453765
- [Background] Villa A, Sankar V, Bassani G, Johnson LB, Sroussi H. Dexamethasone solution and dexamethasone in Mucolox for the treatment of oral lichen planus: a preliminary study. Oral Surg Oral Med Oral Pathol Oral Radiol. 2020 Jun;129(6):585-590. doi: 10.1016/j.oooo.2020.02.014. Epub 2020 Mar 25. PMID 32220595
- [Background] Lavaee F, Shadmanpour M. Comparison of the effect of photodynamic therapy and topical corticosteroid on oral lichen planus lesions. Oral Dis. 2019 Nov;25(8):1954-1963. doi: 10.1111/odi.13188. Epub 2019 Oct 2. PMID 31478283
- [Background] Zhou L, Cao T, Wang Y, Yao H, Du G, Tian Z, Tang G. Clinical observation on the treatment of oral lichen planus with total glucosides of paeony capsule combined with corticosteroids. Int Immunopharmacol. 2016 Jul;36:106-110. doi: 10.1016/j.intimp.2016.03.035. Epub 2016 Apr 26. PMID 27129091